CLINICAL TRIAL: NCT02574949
Title: Impact of Low Frame Rate Fluoroscopy and Cine-angiography on Reducing Operator and Patient Radiation Dose and Impact on Image Quality During Cardiac Catheterization
Brief Title: Impact of Low Frame Rate Fluoroscopy and Cine-angiography on Reducing Operator and Patient Dose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Vladimír Džavík, Director of Research and Innovation-Interventional Cardiology and Coronary Intensive Care Unit, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-8832-AE
Record Dates: First submitted 2015-05-26; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Stable Angina; Unstable Angina; Acute Coronary Syndrome
Keywords: radiation; fluoroscopy; diagnostic
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Acute Coronary Syndrome; Disease | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional rate fluoroscopy (Active Comparator): Radiation: 15 FPS Cine 15 PPS
  Interventions: Radiation: Radiation: 15 FPS Cine 15 PPS
- Intermediate frame rate 7.5 fps (Experimental): Radiation: 7.5 low Frame rate
  Interventions: Radiation: Radiation: 7.5 low Frame rate
- Low frame rate (Experimental): Low Cine 10 PPS
  Interventions: Radiation: Low Cine

INTERVENTIONS:
Radiation: Radiation: 15 FPS Cine 15 PPS — Radiation 15 FPS Cine 15 PPS
  Other Names: Conventional
  Arms: Conventional rate fluoroscopy
Radiation: Radiation: 7.5 low Frame rate — Radiation: Frame rate 7.5 FPS, Cine 15 PPS
  Other Names: Low rate fluoroscopy
  Arms: Intermediate frame rate 7.5 fps
Radiation: Low Cine — Radiation: Frame rate 7.5 FPS, Cine 10 PPS
  Other Names: Low pulse rate Cine
  Arms: Low frame rate

SUMMARY:
The investigators sought to investigate the efficacy of low frame rate (fluoroscopy at 7.5 frames per second (FPS) and Cine at 10 pulse per second (PPS) vs. conventional (15 FPS and 15 PPS) on radiation dose to the patient and the operator during coronary angiography and intervention. In addition, investigators sought to qualitatively assess the effect, if any, of the low frame rate on angiographic image quality.

DETAILED DESCRIPTION:
Minimizing radiation exposure to patient and the operator is considered one of the primary safety concerns in the catheterization laboratory. Patients undergoing diagnostic angiography +/- ad hoc PCI or planned PCI, will be randomised to conventional settings (15 FPS and 15 PPS) or low frame rate settings (7.5 FPS and 15 PPS) or low Cine settings (7.5 FPS and 10 PPS). The patient radiation dose, patient radiation dose area product (DAP), and fluoroscopy time will be measured.

Statistical Analysis:

Demographic and procedural variables will be presented as percentage (categorical variable) or mean ± SD (continuous variable). Patients will be randomized into three arms - a control arm and two intervention arms. The angiographic radiation protocol will adhere to standard practice in both fluoroscopy and cine images at 15 frames/second. The intervention arm will consist of two groups. Group 1 with fluoroscopy images set at 7.5 frames/second and cine images set at 15 frames/second and group 2 with fluoroscopy set at 7.5 frames/second and cine set at 10 frames/second.

Sample size calculations are based on assuming a reduction in radiation dose in group 1 of 10% and in group 2 of 20%. At 5% significance and 80% power, a sample size of 200 patients will be required in each intervention arm. Allowing for a 10% attrition rate, a sample size of 220 patients will be required in each intervention arm with 100 patients in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective or urgent cardiac catheterisation with or without ad-hoc PCI or planned PCI in the pre-specified catheterisation laboratories.

Exclusion Criteria:

* Patients who undergo procedures other than diagnostic coronary angiography or intervention (e.g. electrophysiological procedures).
* Patients participating in other research study requiring higher cine angiography.
* ST-elevation Myocardial Infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Radiation Exposure to patient | During Cardiac catheterization procedure
  Radiation exposure to patient will be measured by Dose-Area product (DAP) collected during the procedure.

SECONDARY OUTCOMES:
Image quality assessment of the coronary angiogram | 12 months
  Coronary angiograms will be assessed by blinded operators for quality of image using a pre-specified tool

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD, FRCPC, Principal Investigator — UHN, Toronto, Canada
Locations (1):
- University Health Network - Peter Munk Cardiac Centre, Toronto, Ontario, Canada